CLINICAL TRIAL: NCT02175654
Title: Phase II Study of Regorafenib as Single Agent for the Treatment of Patients With Metastatic Colorectal Cancer (mCRC) With Any RAS or BRAF Mutation Previously Treated With FOLFOXIRI Plus Bevacizumab
Brief Title: Regorafenib as Single Agent in Patients With Metastatic Colorectal Cancer (mCRC) With Any RAS or BRAF Mutation Previously Treated With FOLFOXIRI Plus Bevacizumab
Acronym: PREVIUM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was prematurely closed due to lack of accrual
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-14-01; 2014-000703-26 (EudraCT Number)
Record Dates: First submitted 2014-06-12; First posted 2014-06-26 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Neoplasms; Metastatic Disease
Keywords: metastatic colorectal cancer; RAS/BRAF mutation; Regorafenib; FOLFOXIRI; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib (Experimental): Regorafenib will be administered orally at the initial dosage of 160 mg per day for 3 weeks, followed by one week of rest, according to the 3/1 regimen
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib

SUMMARY:
The purpose of this study is to assess the efficacy of single-agent regorafenib in the second-line treatment in metastatic colorectal cancer with any RAS or BRAF mutation previously treated with FOLFOXIRI plus bevacizumab in terms of progression-free survival at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the informed consent form.
2. The patient must be able to understand the information and state expressly his or her desire to take part in the study.
3. Age ≥ 18 years.
4. Histologically or cytologically documented adenocarcinoma of the colon or rectum.
5. Patients with metastatic colorectal cancer (stage IV) with any RAS or BRAF mutation.
6. To have received first_line treatment with bevacizumab in combination with chemotherapy with the three drugs 5FU/leucovorin (LV), irinotecan and oxaliplatin (FOLFOXIRI), and

   * have had radiological progression of the disease during the first_line treatment, or
   * have had radiological progression of the disease within a period of ≤ 6 months after the last dose of first-line treatment, or
   * have discontinued part or all of the first_line treatment due to toxicity and have had radiological progression of the disease within a period of ≤ 6 months after the last dose of first-line treatment.

   The patient will have to have received at least one cycle of bevacizumab in combination with FOLFOXIRI + bevacizumab as part of the first_line treatment.

   Patients may have received fluoropyrimidine_based adjuvant treatment with or without oxaliplatin.
7. Existence of at least one measurable unidimensional lesion using CT or MRI based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1
8. Overall Eastern Cooperative Oncology Group (ECOG) performance ≤1.
9. Patient's commitment to compliance with the oral medication throughout the duration of the study
10. Life expectancy of at least 3 months
11. Adequate bone marrow, renal and hepatic function, defined as:

    * Neutrophils ≥ 1500/mm3
    * Platelets ≥100,000/mm3
    * Haemoglobin ≥ 9,0 g/dL
    * Serum Creatinine ≤ 1.5 x LSN
    * Bilirubin levels ≤ 1.5 x LSN
    * AST and ALT levels ≤ 2.5 x ULN (if liver metastases < 5 x ULN)

Exclusion Criteria:

1. Prior treatment with regorafenib.
2. Assignment prior to treatment during this study. Patients who are permanently withdrawn from participation in the study treatment will not be allowed to return to it.
3. Prior or concurrent presence of another neoplastic disease that is different in terms of tumour site and histology of the colorectal cancer in the 5 years prior to the inclusion of the patient in the study, except in situ cervical cancer, superficial bladder carcinoma [Ta (non-invasive), Tis (carcinoma in situ) and T1 (tumour invades lamina propria)] and non-melanoma skin tumours.
4. Presence or history of brain metastases or meningeal tumours.
5. Major surgery, open biopsy or traumatic injury within 28 days prior to the start of patient treatment with the study medication.
6. Extended-field radiotherapy within 4 weeks prior to inclusion or limited-field radiotherapy in the previous 2 weeks. Patients must have recovered from all treatment-related toxicities.
7. Pregnant or breastfeeding women. Women of childbearing age must use adequate contraception. Women of childbearing age must have a negative pregnancy test within 7 days prior to starting with the study medication.
8. Women of childbearing age and men who wish to take part in the study must agree to use adequate contraception from the signing of the informed consent until at least 3 months after stopping the study medication. The investigator or the person designated by him or her will ensure and advise as to the contraceptive methods that should be used.

   Appropriate contraceptive methods include abstinence, oral contraceptives, transdermal patches and injections of sustained-release progestin (starting at least 4 weeks before administration of the IMP), double-barrier method: condom or female condom (diaphragm or cervical/vaginal condom) plus spermicide, intrauterine device (IUD), intrauterine system, implant or vaginal ring (in place at least 4 weeks before administration of the IMP) or male partner sterilisation (vasectomy with documentation of azoospermia) prior to inclusion of the woman in the trial if he is the woman's only sexual partner.
9. Active congestive heart failure class 2 or higher on the New York Heart Association (NYHA) scale.
10. Unstable angina (angina symptoms at rest), new_onset angina (having appeared in the past 3 months) or acute myocardial infarction that has occurred in the 6 months prior to starting with the study medication.
11. Cardiac arrhythmias that require anti-arrhythmic therapy (only beta blockers and digoxin would be allowed as concomitant medication for these patients).
12. Uncontrolled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg) despite proper medical management.
13. Patients with phaeochromocytoma.
14. Pleural effusion or ascites that cause breathing difficulties (dyspnoea of grade ≥ 2 of the CTC).
15. Venous or arterial thromboembolism or embolic events such as cerebrovascular accidents (including transient ischaemic attacks), deep vein thrombosis or pulmonary thromboembolism that have occurred in the 6 months prior to starting with the study medication.
16. Active infection > grade 2 based on the NCI CTC, v. 4.0.
17. Human immunodeficiency virus (HIV) infection.
18. Active hepatitis B or C, or hepatitis B or C infection that requires treatment with antiviral drugs.
19. Patients with mental disorders that require medication.
20. History of organ transplants.
21. Patients with evidence or history of bleeding diathesis. Any bleeding or bleeding event > Common Toxicity Criteria for Adverse Effects (CTCAE) grade 3 in the 4 weeks prior to starting with the study medication.
22. Presence of unhealed wounds, ulcers or bone fractures.
23. Kidney failure requiring haemodialysis or peritoneal dialysis.
24. Dehydration based on NCI CTC criteria, version 4, of > 1.
25. Substance abuse or a history of medical, social or psychological conditions that may interfere with study participation or compliance with the efficacy and safety assessments planned in the study.
26. Known hypersensitivity to regorafenib or any of its excipients.
27. Presence of any disease or medical condition that might interfere with patient safety or may compromise treatment compliance with it.
28. Interstitial lung disease with signs and symptoms present at the time of signing the informed consent.
29. Patients who are unable to swallow oral medication.
30. Persistent proteinuria > grade 3 based on the NCI CTC, version 4.0 (> 3.5 g/24 hours).
31. Intestinal malabsorption syndrome.
32. Close personal relationship with the research staff, such as family members of the investigator or dependents (e.g. employees or students of the research centre).
33. Unresolved toxicity grade > 1 based on the NCI CTC, version 4.0 (except alopecia), related to any previous therapy or procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate at 6 months | 6 months

SECONDARY OUTCOMES:
Objective response rate based on the Response Evaluation Criteria in Solid Tumors criteria | 36 months
Disease control rate | 36 months
Response according other criteria (Appendix 9) | 36 months
Time to response | 36 months
Progression free survival | 36 months
Time to treatment failure | 36 months
Response duration | 36 months
Duration of stable disease | 36 months
Overall survival | 36 months
Time to progression | 36 months
Incidence and severity of adverse events (AE) (NCI CTC, version 3.0) | 36 months
Changes in laboratory values | baseline and end of treatment, an expected average of 4 months
  hemoglobin, hematocrit, platelets, creatinine, total bilirubin, alkaline phosphatase, ALT, AST, BUN or urea, glucose, sodium, potassium, calcium, phosphorus, LDH, GGT, magnesium, albumin, total protein, uric acid and lipase.
Change in vital signs (weight loss and hypertension) | baseline and end of treatment, an expected average of 4 months
Incidence of dose adjustments and compliance | 36 months
Incidence of concomitant medication | 36 months
Changes in ECOG performance status over time from baseline | baseline and end of treatment, an expected average of 4 months

OTHER OUTCOMES:
microRNA expression level in the Peripheral Blood | 36 months
Biomarkers associated with cell and tumour growth and/or the mechanism of action of regorafenib and their correlation with patients' clinical progression for efficacy and safety parameters. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Pilar García Alfonso, MD, Study Chair — Gregorio Marañón Hospital; Manuel Benavides, MD PhD, Study Chair — Regional Universitario Hospital
Locations (1):
- Spanish Cooperative Group for Digestive Tumour Therapy (TTD), Madrid, Spain

REFERENCES:
- [Derived] Garcia-Alfonso P, Benavides M, Falco E, Munoz A, Gomez A, Sastre J, Rivera F, Montagut C, Salgado M, Lopez-Ladron A, Lopez R, Ruiz de Mena I, Duran G, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumors (TTD). Single-Agent Regorafenib in Metastatic Colorectal Cancer Patients with Any RAS or BRAF Mutation Previously Treated with FOLFOXIRI plus Bevacizumab (PREVIUM Trial). Oncologist. 2018 Nov;23(11):1271-e128. doi: 10.1634/theoncologist.2018-0316. Epub 2018 Aug 17. PMID 30120161
- See also: Related Info — http://www.ttdgroup.org